CLINICAL TRIAL: NCT01005654
Title: Prospective Comprehensive Molecular Analysis of Endocrine Neoplasms
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090242; 09-C-0242
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-08

CONDITIONS: Endocrine Tumors; Thyroid Neoplasms; Parathyroid Neoplasms; Adrenal Neoplasm; Neuroblastoma
Keywords: Gene Expression; Epigenetic (methylation); Tissues Histological Evaluations; Establishment of Tumor Cell Lines; Metabolite and Protein Expression; Natural History; Adrenal Cancer; Endocrine Tumor; Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms; Parathyroid Neoplasms; Adrenal Gland Neoplasms; Neuroblastoma; Endocrine Gland Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/ Cohort 1: Participants with endocrine neoplasm or pre or potentially malignant condition of the endocrine system, scheduled to have surgery or biopsy

SUMMARY:
Background:

* Endocrine neoplasms (tumors) are among the fastest growing tumors in incidence in the United States. Furthermore, it is often difficult to distinguish between benign or malignant tumors in cancers of the thyroid, parathyroid, adrenal gland, and pancreas. More research is needed to improve detection and treatment options for patients who develop these kinds of cancer.
* Researchers are interested in studying the molecular changes that are involved in endocrine cancer development and growth. To collect a sample of tumor specimens and healthy tissue for further study, researchers are specifically looking for samples from participants who are scheduled for surgery or biopsy on endocrine tumors.

Objectives:

- To collect samples of precancerous, cancerous, and healthy tissue from individuals who are scheduled for surgery or biopsy of endocrine system tumors.

Eligibility:

- Individuals who have a tumor in or around their thyroid, parathyroid, adrenal gland, pancreas, or any neuroendocrine tissue, and are scheduled for surgery at the National Institutes of Health Clinical Center.

Design:

* Participants in this study will provide blood and urine samples prior to surgery.
* During the surgery or biopsy, pieces of the tumor or precancerous growth and pieces of normal tissue near to the tumor will be removed for ongoing and future research. The rest of the tumor or growth will be sent for analysis.
* After surgery, participants will receive routine care until discharge, and doctors will discuss possible treatment options. If there is an appropriate NIH protocol, participants may choose to be treated at the NIH.
* After discharge, participants will return to the clinic for a routine postoperative check about 6 weeks following the operation, and then may be followed yearly at the Clinical Center or by phone....

DETAILED DESCRIPTION:
Background:

Endocrine neoplasms are among the fastest growing tumors in incidence in the United States. Between 1995 and 2005, the incidence of thyroid carcinoma has increased 98 percent.

Tumors of the thyroid, parathyroid, adrenal gland and gastrointestinal-pancreatic neuroendocrine tumors are among some of the most difficult tumors to clinically and histopathological distinguish as benign or malignant.

Moreover, endocrine neoplasms provide an extremely important model for studying the important molecular changes that lead to carcinogenesis because of their diverse clinical behavior, even when having the same TNM stage and histologic features.

The Surgical Oncology Program (formerly known as Endocrine Oncology Branch), NCI has a focus on studying the molecular changes that are involved in endocrine cancer initiation and progression. In addition, this section has primary responsibility for providing endocrine surgery consultative services to the NIH. As such, we are uniquely positioned to acquire and perform important studies to help identify diagnostic and predictive markers as well as therapeutic targets that may have significant clinical ramifications.

Objectives:

To develop a genetic, epigenetic, metabolomic, and proteomic profile of endocrine neoplasm that will allow us to distinguish benign from malignant tumor for each of the endocrine histologies under study. This objective will drive the statistical endpoints of the study.

Eligibility:

Participants with radiographic evidence of, biochemical evidence of, or histologically/cytologically proven, endocrine neoplasms, including lesions of the thyroid, parathyroid, adrenal, extra-adrenal endocrine nests, paragangliomas, neuroblastomas, pancreas and gastrointestinal tract. Or participants with a described pre or potentially malignant condition that requires surgery or biopsy as a part of the standard of care treatment and/or follow up.

Participants must have an ECOG performance score of 0-2.

Participants must have physical examination parameters within acceptable limits by standard of practice guidelines prior to biopsy or surgery.

Design:

A tissue acquisition trial in which tissues will be obtained at the time of surgical operation for the removal of neoplasms of the thyroid, parathyroid, adrenal, pancreas, paragangliomas and/or extra adrenal nests of neuroendocrine tissue, and gastrointestinal neuroendocrine tumors.

At the time of surgical operation, blood samples will be obtained from the operative field during the removal of neoplasms of the thyroid, parathyroid, adrenal, pancreas, paragangliomas and/or extra adrenal neuroendocrine tissue and gastrointestinal neuroendocrine tumors.

No investigational therapy will be given.

It is anticipated that 2,300 participants will be followed on this study, however, to account for screening up to 2,415 participants may be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants who have an endocrine neoplasm based on radiographic and biochemical testing, or histologically/cytologically proven lesions of the thyroid, parathyroid, adrenal, extra-adrenal endocrine nests, paragangliomas, neuroblastomas, gastrointestinal

track and pancreas or participants with a described pre or potentially malignant condition that requires surgery or biopsy as a part of the standard of care treatment and/or follow up.

* Participants referred to the Endocrine Consult Service on other protocols for surgical evaluation of endocrine disorders based on radiographic and biochemical testing, or histologically/cytologically proven lesions of the thyroid, parathyroid, adrenal, extra-adrenal endocrine nests, paragangliomas, neuroblastomas and pancreas.
* Participants must have an ECOG performance score of 0-2.
* Participants must have physical examination parameters within acceptable limits by standard of practice guidelines prior to biopsy or surgery.
* Participants must be planning to undergo surgery or biopsy as part of their treatment plan. Note: Participants will not be enrolled exclusively for the procurement of tissue samples.
* Age >= 4 years of age.

EXCLUSION CRITERIA:

None.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary clinical@@@
Sampling Method: Non-Probability Sample
Enrollment: 2415 (Estimated)
Dates: Start 2009-10-07 (Actual)

PRIMARY OUTCOMES:
To develop a genetic, epigenetic, metabolomic, and proteomic profile of endocrine neoplasm that will allow us to distinguish benign from malignant tumor for each of the endocrine histologies under study. | 10 years
  To develop a genetic, epigenetic, metabolomic, and proteomic profile of endocrine neoplasm that will allow us to distinguish benign from malignant tumor for each of the endocrine histologies under study.

SECONDARY OUTCOMES:
To utilize the tissue obtained from these endocrine neoplasms for studies of gene expression, epigenetic (methylation) changes, and metabolite and protein expression. | at the time of procedure or biopsy
  Obtained endocrine neoplasm tissue will be used for studies of gene expression, epigenetic (methylation) changes, and metabolite and protein expression.
To obtain, when accessible, normal endocrine and other adjacent tissue for comparison with the neoplastic tissue including the comparison of genomic profiling data to determine the best approach for normalizing expression data. | at the time of procedure or biopsy
  When accessible, normal endocrine and other adjacent tissue will be obtained for comparison with the neoplastic tissue for genomic profiling to determine the best approach for normalizing expression data.
To collect tissues from endocrine neoplasms arising in the thyroid, parathyroid, adrenal, pancreas, extra-adrenal neuroendocrine nests, and gastrointestinal neuroendocrine tumors for future analysis and correlation with clinical outcome. | at the time of procedure or biopsy
  Obtained endocrine neoplasm tissue in the thyroid, parathyroid, adrenal, pancreas, extra-adrenal neuroendocrine nests, and gastrointestinal neuroendocrine tumors will be collected for future analysis and correlation with patient clinical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Naris Nilubol, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Smigal C, Thun MJ. Cancer statistics, 2006. CA Cancer J Clin. 2006 Mar-Apr;56(2):106-30. doi: 10.3322/canjclin.56.2.106. PMID 16514137
- [Background] Lee PK, Jarosek SL, Virnig BA, Evasovich M, Tuttle TM. Trends in the incidence and treatment of parathyroid cancer in the United States. Cancer. 2007 May 1;109(9):1736-41. doi: 10.1002/cncr.22599. PMID 17372919
- [Background] Howlett DC, Speirs A. The thyroid incidentaloma--ignore or investigate? J Ultrasound Med. 2007 Oct;26(10):1367-71. doi: 10.7863/jum.2007.26.10.1367. PMID 17901140
- [Derived] Neychev V, Steinberg SM, Yang L, Mehta A, Nilubol N, Keil MF, Nieman L, Stratakis CA, Kebebew E. Long-Term Outcome of Bilateral Laparoscopic Adrenalectomy Measured by Disease-Specific Questionnaire in a Unique Group of Patients with Cushing's Syndrome. Ann Surg Oncol. 2015 Dec;22 Suppl 3(Suppl 3):S699-706. doi: 10.1245/s10434-015-4605-1. Epub 2015 May 13. PMID 25968622
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2009-C-0242.html